CLINICAL TRIAL: NCT07160569
Title: Microbiological and Clinical Characteristics of Severe Infections Caused by Carbapenem-Resistant Enterobacterales: A Prospective Multicenter Study in Southern Italy (the MICE Study)
Brief Title: Microbiological and Clinical Characteristics of Severe Infections Caused by Carbapenem-Resistant Enterobacterales
Acronym: MICE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID7409
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Treatment group-ceftazidime/avibactam: 30 patients receiving this treatment, isolation of CRE from a clinically relevant sample considered to be the site of infection: pneumonia, UTI, IAI, spondylodiscitis and BSI.
  Interventions: Diagnostic Test: Whole Genome Sequencing (WGS), Sequence Type Analysis (ST)
- Treatment group-meropenem/vaborbactam: 30 patients receiving this treatment, isolation of CRE from a clinically relevant sample considered to be the site of infection: pneumonia, UTI, IAI, spondylodiscitis and BSI.
  Interventions: Diagnostic Test: Whole Genome Sequencing (WGS), Sequence Type Analysis (ST)
- Treatment group-cefiderocol: 30 patients receiving this treatment, isolation of CRE from a clinically relevant sample considered to be the site of infection: pneumonia, UTI, IAI, spondylodiscitis and BSI.
  Interventions: Diagnostic Test: Whole Genome Sequencing (WGS), Sequence Type Analysis (ST)

INTERVENTIONS:
Diagnostic Test: Whole Genome Sequencing (WGS), Sequence Type Analysis (ST) — Whole Genome Sequencing (WGS), Sequence Type Analysis (ST), resistome, viruloma, and phenotypic resistance of CRE
  Other Names: Whole Genome Sequencing (WGS), Sequence Type Analysis (ST), resistome, viruloma, and phenotypic resistance of CRE

SUMMARY:
Severe infections caused by carbapenem-resistant Enterobacterales (CRE) represent a challenge for the clinicians, considering the high mortality rate of these infections. Data regarding the prevalence of CRE, clonal analysis, resistant genes (resistome) and virulence genes (virulome) molecular analyses, and clinical outcomes of infected patients are scarce. Thus, creating a network to Standardize and implement microbiological sourveillance could be crucial to answer this challenge. Our group consisting of the, UOC of Infectious Diseases and UOC of Microbiology (Prof Sanguinetti), the Microbiology Unit of the University of Catania (Prof. Stefania Stefani), the local Infectious Disease Unit (Dr Carmelo Iacobello) the Microbiology Unit of the "Magna Graecia'' University (Prof. Giovanni Matera) and the UOC of Infectious and Tropical Diseases UMG Catanzaro Prof Enrico Maria Trecarichi, has already started a project with promising ad interim results on this topic.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. isolation of CRE from a clinically relevant sample considered to be the site of infection: pneumonia, UTI, IAI, spondylodiscitis and BSI.
3. Patients who by clinical practice have received at least one dose of the following drugs from ceftazidime-avibactam, meropenem-vaborbactam, and cefiderocol.
4. Signature of Informed Consent

Exclusion Criteria:

1. Subjects under 18 years of age
2. absence of CRE infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with confirmed CRE infections, defined as pathogens resistant to meropenem, ertapenem, and imipenem, assessed by EUCAST (European Committee on Antimicrobial Susceptibility Testing) and who have received at least one dose of the following drugs: ceftazidime-avibactam, meropenem-vaborbactam, and cefiderocol.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of the susceptibility/resistance | 12 months
  prevalence of the susceptibility/resistance patterns of ceftazidime- avibactam, meropenem-vaborbactam and cefiderocol in all the CRE isolates

SECONDARY OUTCOMES:
Prevalence of different Sequence Type Analysis | 12months
  To assess the prevalence of different Sequence Type Analysis (ST), resistome and virulome of the collected CRE isolates
Odds ratio for the association between multiple factors | 12 months
  To assess the odds ratio for the association of the primary endpoint with demographic, clinical, and therapeutic factors

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Torti, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (4):
- Italy (4):
  - Fondazione Policlinico Universtiario Agostino Gemelli IRCCS, Rome, Roma
  - Unit of Infectious and Tropical Diseases, Azienda Ospedaliera "Cannizzaro", Catania, Catania
  - Unit of Infectious and Tropical Diseases, University "Magna Graecia", Catanzaro, Catanzaro
  - Unit of Infectious and Tropical Diseases, Azienda Ospedaliera "Bianchi-Melacrino-Morelli", Reggio Calabria, Reggio Calabria

IPD SHARING:
Plan to Share IPD: No